CLINICAL TRIAL: NCT01655225
Title: A Phase 1 First-in-Human Dose Study of LY3023414 in Patients With Advanced Cancer
Brief Title: A Study of LY3023414 in Participants With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13517; I6A-MC-CBBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-19; First posted 2012-08-01 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Advanced Cancer; Metastatic Cancer; Non-Hodgkin's Lymphoma; Metastatic Breast Cancer; Malignant Mesothelioma; Non-small Cell Lung Cancer
Keywords: Advanced Breast Cancer; Advanced Lung Cancer; Mesothelioma; Lymphoma
MeSH Terms: conditions — Neoplasm Metastasis; Lymphoma, Non-Hodgkin; Breast Neoplasms; Mesothelioma, Malignant; Carcinoma, Non-Small-Cell Lung; Mesothelioma; Lymphoma | interventions — LY3023414; Midazolam; Fulvestrant; Pemetrexed; Cisplatin; abemaciclib; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (9):
- Part A: LY3023414 Once Daily (Experimental): LY3023414 administered orally once daily (QD) at escalating doses for two 21 day cycles to participants with advanced/metastatic cancer (including lymphoma); participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414
- Part A2: LY3023414 Twice Daily (Experimental): LY3023414 administered orally twice daily (BID) at escalating doses for two 21 day cycles to participants with advanced/metastatic cancer (including lymphoma); participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414
- Part B1 : LY3023414 + Midazolam (Experimental): LY3023414 administered orally BID for two 21 day cycles to participants with advanced/metastatic cancer; participants receiving benefit may continue until disease progression or discontinuation. Dose based on Part A. 0.2 milligrams (mg) midazolam administered orally once before LY3023414 on Day 1 and once after LY3023414 on Day 15.
  Interventions: Drug: LY3023414; Drug: Midazolam
- Part B2: LY3023414 + Fulvestrant (Experimental): LY3023414 administered orally BID for two 28 day cycles to participants with advanced/metastatic breast cancer; participants receiving benefit may continue until disease progression or discontinuation. 500 mg fulvestrant administered IM once every 28 days.
  Interventions: Drug: LY3023414; Drug: Fulvestrant
- Part B3: LY3023414 (Experimental): LY3023414 administered orally BID for two 21 day cycles to participants with malignant mesothelioma; participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414
- Part B4: LY3023414 + pemetrexed/cisplatin (Experimental): LY3023414 administered orally BID for two 21 day cycles to participants with malignant mesothelioma; participants receiving benefit may continue until disease progression or discontinuation. 500 mg/m2 pemetrexed and 75 mg/m2 administered IV once every 21 days.
  Interventions: Drug: LY3023414; Drug: Pemetrexed; Drug: Cisplatin
- Part B5: LY3023414 (Experimental): LY3023414 administered orally BID for two 21 day cycles to participants with indolent non-Hodgkin's lymphoma; participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414
- Part B6: LY3023414 (Experimental): LY3023414 administered orally BID for two 21 day cycles to participants with squamous NSCLC; participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414
- Part B7: LY3023414 + Abemaciclib + Letrozole (Experimental): LY3023414 administered orally BID with abemaciclib administered orally BID and letrozole administered orally once a day for two 28 day cycles to participants with breast cancer; participants receiving benefit may continue until disease progression or discontinuation.
  Interventions: Drug: LY3023414; Drug: Abemaciclib; Drug: Letrozole

INTERVENTIONS:
Drug: LY3023414 — Administered orally. Dose of 20 to 600 mg, as determined in Part A.
Drug: Midazolam — 0.2 mg administered orally once before LY3023414 on Day 1 and once after LY3023414 on Day 15.
  Arms: Part B1 : LY3023414 + Midazolam
Drug: Fulvestrant — 500 mg administered IM on Day 1 and Day 15 in cycle 1 and Day 1 every 28 days for additional cycles.
  Arms: Part B2: LY3023414 + Fulvestrant
Drug: Pemetrexed — 500 mg/m2 administered IV once on Day 1 every 21 days
  Other Names: Alimta
  Arms: Part B4: LY3023414 + pemetrexed/cisplatin
Drug: Cisplatin — 75 mg/m2 administered IV once on Day 1 every 21 days
  Arms: Part B4: LY3023414 + pemetrexed/cisplatin
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219
  Arms: Part B7: LY3023414 + Abemaciclib + Letrozole
Drug: Letrozole — Administered orally
  Arms: Part B7: LY3023414 + Abemaciclib + Letrozole

SUMMARY:
The purpose of this study is to find a recommended dose level and schedule of dosing LY3023414 that can safely be taken by participants with advanced or metastatic cancer. The study will also explore the changes to various markers in blood cells and potentially tumor cells. Finally, the study will help document any antitumor activity this drug may have.

In Part A of this study, participants with advanced/metastatic cancer (including lymphoma) will receive increasing doses of LY3023414. In Part B, LY3023414 will be explored in different types of cancer, including breast and lung cancer, lymphoma and mesothelioma.

ELIGIBILITY:
Inclusion Criteria:

* Parts A, A2 & B1: Participants must have pathological evidence of a diagnosis of advanced and/or metastatic cancer and must be, in the judgment of the investigator, an appropriate candidate for experimental therapy
* Part B2: Participants must have advanced, recurrent, or metastatic breast cancer that is refractory to aromatase inhibitors (AI) with either disease recurrence or disease progression; must be hormone receptor positive (HR+) and human epidermal growth factor receptor 2 (HER2)-negative; must be of postmenopausal status or beginning ovarian suppression with a luteinizing hormone-releasing hormone (LHRH) agonist
* Part B3 only: Participants must have malignant pleural or peritoneal mesothelioma
* Part B4 only: Participants must have malignant pleural or peritoneal mesothelioma and appropriate candidate for treatment with cisplatin/pemetrexed; no prior systemic chemotherapy
* Part B5 only: Participants must have histologically confirmed diagnosis of B-cell iNHL, with histological subtype; prior treatment with ≥2 prior chemotherapy- or immunotherapy-based regimens for iNHL
* Part B6 only: Participants must have squamous NSCLC; documented evidence of an activating molecular aberration of the PI3K/mTOR pathway
* Parts B2, B3 & B6 only: Must have adequate tumor tissue sample from archival biopsy available, or willingness to undergo a fresh tumor biopsy
* Parts B3, B4, B5 & B6: No previous treatment with any PI3K and/or mTOR inhibitor
* Part B7: Must have a diagnosis of HR+ and HER2- breast cancer; have locoregionally recurrent disease not amenable to resection or radiation therapy with curative intent or metastatic disease; no previous treatment or currently receiving 1 of the following treatments for locoregionally recurrent or metastatic breast cancer (chemotherapy, endocrine therapy, CDK4/6 inhibitor, and PI3K and/or mTOR inhibitor)
* Measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1), modified RECIST or Revised Response Criteria for Malignant Lymphoma
* Have adequate organ function, including: Absolute neutrophil count (ANC) at least 1.5 x 109/Liter (L), platelets at least 100 x 109/L, and hemoglobin at least 8 grams/deciliter (g/dL); bilirubin no more than 1.5 times upper limits of normal; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) no more than 2.0 times upper limits of normal; Serum creatinine no more than 1.5 times upper limits of normal or calculated creatinine clearance >45 milliliters/minute (mL/min)
* Have a performance status of at least 1 on the Eastern Cooperative Oncology Group (ECOG) scale and life expectancy >6 months
* Have discontinued all previous cancer therapies (except nonsteroidal aromatase inhibitors for participants in Part B2), and any agents that have not received regulatory approval for any indication, for at least 21 days or 5 half lives prior to study enrollment, whichever is shorter, and recovered from the acute effects of therapy. Participants must have discontinued mitomycin-C or nitrosourea therapy for at least 42 days
* Are able to swallow capsules

Exclusion Criteria:

* Have serious preexisting medical conditions
* Have symptomatic central nervous system (CNS) malignancy (with the exception of medulloblastoma) or metastasis (screening not required).
* Have known acute or chronic leukemia or current hematologic malignancies (except iNHL for patients in Part B5) that, in the judgment of the investigator and sponsor, may affect the interpretation of results
* Have an active fungal, bacterial, and/or known viral infection
* Have a second primary malignancy that in the judgment of the investigator and sponsor may affect the interpretation of results (Part B only)
* Part B1 only: No concomitant medications that are strong inhibitors or inducers of cytochrome P450 3A4 (CYP3A4) or midazolam
* Intolerance to any previous treatment with any phosphatidylinositol-3-kinase (PI3K) and/or mammalian target of rapamycin (mTOR) inhibitor.
* Participants with active alcohol abuse, as determined by the investigator
* Have a history of New York Heart Association (NYHA) Class ≥3, unstable angina, or myocardial infarction (MI) in 6 months prior to study drug administration
* Have QT corrected interval of >450 milliseconds (msec) on screening electrocardiogram (ECG)
* Have insulin-dependent diabetes mellitus or a history of gestational diabetes mellitus.
* Part B only: Hypersensitivity to study drugs given in combination with LY3023414

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 dose | Baseline to disease progression or participant discontinuation (estimated 9 weeks)

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum concentration (Cmax) | Predose up to 12 hours postdose
Pharmacokinetics: Time of maximal concentration | Predose up to 12 hours postdose
Number of participants with tumor response | Baseline to disease progression or participant discontinuation (estimated 9 weeks)
Potential of LY3023414 to inhibit CYP3A4-mediated metabolism | Baseline through Cycle 1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Peggy and Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
- Azienda Ospedaliero - Universitaria S. Luigi Gonzaga, Orbassano, Torino, Italy
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico

REFERENCES:
- [Derived] Zauderer MG, Alley EW, Bendell J, Capelletto E, Bauer TM, Callies S, Szpurka AM, Kang S, Willard MD, Wacheck V, Varghese AM. Phase 1 cohort expansion study of LY3023414, a dual PI3K/mTOR inhibitor, in patients with advanced mesothelioma. Invest New Drugs. 2021 Aug;39(4):1081-1088. doi: 10.1007/s10637-021-01086-6. Epub 2021 Mar 4. PMID 33660194
- See also: A Study of LY3023414 in Participants With Advanced Cancer — https://trials.lillytrialguide.com/en-US/trial/1hEgh09hSQ64QyAaacI6my